CLINICAL TRIAL: NCT07136064
Title: Jockey Club Support Project to Enhance Emotion Regulation Skills and Resilience of Cross-Boundary Families: A Randomized Controlled Trial
Brief Title: Jockey Club Support Project
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other); International Social Services Hong Kong Branch (Unknown)
Responsible Party: Principal Investigator, Dr. Nancy Xiaonan Yu, Professor, City University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Jockey Club Support Project
Record Dates: First submitted 2025-08-13; First posted 2025-08-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Family Relations; Resilience; Emotion Regulation
Keywords: cross-boundary families; resilience; emotion regulation; randomized controlled trial
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): This arm will receive training in emotion regulation skills, including mindfulness skills to help redeploy their attention, cognitive reappraisal skills to analyze stimuli or emotion-eliciting events from a more comprehensive perspective, situation change skills to regulate emotions by exposing oneself to nature, experiential acceptance skills through metaphor, and breathing techniques. They will also receive training in theories of the family emotion system.
  Interventions: Behavioral: Emotion Regulation Skills Training
- Control (Active Comparator): This arm will be trained to moderate their and their family members' use of commercial electronics. They will do so by learning mechanisms behind addictions, family communication skills, and various substitute activities for commercial electronics usage.
  Interventions: Behavioral: Moderation in Consumer Electronics Use Training

INTERVENTIONS:
Behavioral: Emotion Regulation Skills Training — This arm will receive training in emotion regulation skills, including mindfulness skills to help redeploy their attention, cognitive reappraisal skills to analyze stimuli or emotion-eliciting events from a more comprehensive perspective, situation change skills to regulate emotions by exposing oneself to nature, experiential acceptance skills through metaphor, and breathing techniques. They will also receive training in theories of the family emotion system.
  Arms: Intervention Arm
Behavioral: Moderation in Consumer Electronics Use Training — This arm will be trained to moderate their and their family members' use of commercial electronics. They will do so by learning mechanisms behind addictions, family communication skills, and various substitute activities for commercial electronics usage.
  Arms: Control

SUMMARY:
Guided by the process model of emotion regulation, integrative affect-regulation framework for resilience, and the reciprocal dynamics of emotion, affect, and resilience in the family system, researchers will develop a parallel intervention to incorporate two key members in Mainland-Hong Kong cross-boundary families: a parent and a child by improving their affect/emotion regulation skills, de-escalate family conflicts, and flourish under hardships. Specifically, researchers predict that participants in the intervention group will report greater improvement in resilience, emotion regulation, psychological well-being, family harmony, and social connectedness than those in the control group.

DETAILED DESCRIPTION:
Researchers will conduct a randomized controlled trial (RCT) intervention study targeting cross-boundary families' affect/emotion regulation skills as well as personal and family resilience. Researchers will implement two arms with the allocation ratio of 2:1. As most cross-boundary children are preoccupied with after-school academies and extracurricular activities, participating parents will receive four group activity sessions, while children will receive two sessions. The intervention themes and skills are the same for parents and children but condensed for children.

Researchers will collaborate with the International Social Services Hong Kong Branch (Shenzhen) (hereinafter referred to as "ISS"), an NGO that has served cross-boundary families in Shenzhen for over 30 years.

ELIGIBILITY:
Inclusion Criteria for Parents:

1. have at least one child between the fifth and twelfth grade;
2. can participate in the intervention with their child;
3. are Hong Kong residents or have a family member who is a Hong Kong resident;
4. live in Shenzhen.

Inclusion Criteria for Children:

1. are between the fifth and twelfth grade;
2. are Hong Kong residents or have a family member who is a Hong Kong resident;
3. live in Shenzhen.

Exclusion Criteria:

(a) those who have current diagnoses of severe physical or mental illnesses;

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Resilience | Baseline, 4 weeks, 8 weeks
  Participants' psychological resilience will be measured by the 25-item Connor-Davidson Resilience Scale. Participants will report their perceived psychological resilience of self on a 5-point Likert scale (0 = strongly disagree; 4 = strongly agree). Higher total scores indicate higher levels of psychological resilience.
Cognitive Emotion Regulation | Baseline, 4 weeks, 8 weeks
  Participants' use of adaptive cognitive emotion regulation strategies will be measured by corresponding subscales of the Cognitive Emotion Regulation Questionnaire (CERQ). The study will employ five subscales, including acceptance, positive refocusing, refocus on planning, positive reappraisal, and putting into perspective, as these strategies are the targets of the intervention. Each subscale includes four items. Participants will report their use of each strategy on a 5-point Likert scale (1 = almost never; 5 = almost always). Higher scores for each subscale indicate more use of the corresponding cognitive emotion regulation strategy.
Behavioral Emotion Regulation | Baseline, 4 weeks, 8 weeks
  Participants' use of adaptive behavioral emotion regulation strategies will be measured by corresponding subscales of the Behavioral Emotion Regulation Questionnaire (BERQ). The study will employ two subscales (seeking distraction and putting into perspective) as these strategies are the targets of the intervention. Each subscale includes four items. Participants will report their use of each strategy on a 5-point Likert scale (1 = almost never; 5 = almost always). Higher scores for each subscale indicate more use of the corresponding behavioral emotion regulation strategy.
Affective Experiences | Baseline, 4 weeks, 8 weeks
  Participants' affective experiences will be measured by the International Positive and Negative Affect Schedule Short Form (I-PANAS-SF). Participants will report their experienced positive and negative affect on a 10-item, 5-point Likert scale (1 = never; 5 = always). Higher scores indicate higher levels of positive or negative affect.
Depression and Anxiety Symptoms | Baseline, 4 weeks, 8 weeks
  Participants' depression and anxiety symptoms will be measured by the Patient Health Questionnaire (PHQ-4). On this 4-point Likert scale from 0 to 3, participants will report their frequency of depression and anxiety symptoms. Higher scores indicate more severe symptoms.
Well-being | Baseline, 4 weeks, 8 weeks
  Participants will also complete the 5-item WHO Well-Being Index (WHO-5). They will report their well-being with a 6-point Likert scale (0 = at no time; 5 = all of the time). Higher scores indicate higher levels of well-being.

SECONDARY OUTCOMES:
Family Resilience | Baseline, 4 weeks, 8 weeks
  Participants' family resilience will be measured by the Walsh Family Resilience Questionnaire Short Version (WFRQ-9). Participants will report their perceived family resilience on a 5-point Likert scale (1 = rarely/never; 5 = almost always), with higher scores indicating higher levels of family resilience.
Family harmony | Baseline, 4 weeks, 8 weeks
  Participants will complete the 8-item Family Harmony Scale. Participants will report their perceived level of family harmony on this 8-item, 5-point Likert scale (1 = strongly disagree; 5 = strongly agree). Higher scores indicate higher levels of family harmony.
Parent-Child Conflicts | Baseline, 4 weeks, 8 weeks
  Participants' recent conflicts with their children or parents will be measured by two single-item scales. Participants will report their frequency of conflicts on one scale and the intensity on another. Each scale ranges from one (no conflicts) to five (four or more times of conflicts or very severe conflicts).
Parenting Self-Efficacy | Baseline, 4 weeks, 8 weeks
  Parents will report their parenting self-efficacy on the Parenting Sense of Competence Scale. Participants will indicate their perceived self-efficacy in parenting activities on a 17-item, 6-point Likert scale (1 = strongly disagree; 6 = strongly agree). Higher scores indicate higher levels of self-efficacy in parenting.
Parental Stress | Baseline, 4 weeks, 8 weeks
  Parents will complete the Parental Stress Scale (PSS) to measure their subjective feelings of stress as a parent. Participants will report their perceived parental stress on a 18-item, 6-point Likert scale (1 = strongly disagree; 6 = strongly agree). Higher scores indicate higher levels of parental stress.

OTHER OUTCOMES:
Sense of Community | Baseline, 4 weeks, 8 weeks
  Participants will report their sense of community on the Brief Sense of Community Scale (BSCS). The measurement includes four subscales: needs fulfillment, group membership, influence, and shared emotional connection. Participants will report their perceived sense of community of self on a 5-point Likert scale (1 = strongly disagree; 5 = strongly agree). Higher scores indicate participants' higher sense of community.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy X Yu, Doctoral, Principal Investigator — City University of Hong Kong
Locations (1):
- International Social Service Hong Kong Branch, Shenzhen, Guangdong, China